CLINICAL TRIAL: NCT01717352
Title: Increasing Sleep Duration: A Novel Approach to Weight Control. Study 5-Randomized Trial of Sleep Plus Eating Routines as An Approach to Prepare Participants for Weight Loss
Brief Title: Sleep Plus Eating Routines for Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Professor of Psychiatry & Human Behavior, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01CA150387-Study 5; U01CA150387 (NIH)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Overweight and Obesity
Keywords: Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Loss Education (Active Comparator): Provides participants with important information about weight control and healthy eating prior to treatment to prepare participants for participation in a weight loss program and enhance outcomes.
  Interventions: Behavioral: Weight Loss Education
- Sleep and Eating Routine (Active Comparator): Establish a consistent sleep and eating routine prior to treatment to prepare participants for participation in a weight loss program and enhance outcomes.
  Interventions: Behavioral: Sleep and Eating Routine

INTERVENTIONS:
Behavioral: Weight Loss Education
  Arms: Weight Loss Education
Behavioral: Sleep and Eating Routine
  Arms: Sleep and Eating Routine

SUMMARY:
The present study will test the effectiveness of two different approaches for preparing overweight/obese individuals for weight loss: 1)providing important information about weight control, including dispelling common myths; or 2) developing a consistent sleep and eating routine to prepare for the challenges of a weight control intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 21 to 65
* BMI 25 to 45
* sleep 7 hours or less most nights

Exclusion Criteria:

* use of medications affecting sleep
* sleep apnea
* shift work

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Weight | 20 weeks

SECONDARY OUTCOMES:
Executive Control | 4 and 20 weeks
  Executive control is measured by a variety of computer assessments. These include Go-No Go, delayed discounting, and perseverence as measured by mirror tracing and a hand grip task.

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States